CLINICAL TRIAL: NCT05387252
Title: Dose-response Study a Glucoside- and Rutinoside-rich Crude Material in Relieving Side Effects of COVID-19 Vaccines
Brief Title: Glucoside- and Rutinoside-rich Crude Material for Relieving Side Effects of COVID-19 Vaccines
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, El-Wui Loh, Associate Professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: N202202030
Record Dates: First submitted 2022-05-19; First posted 2022-05-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Vaccine Adverse Reaction; Side-Effect
Keywords: COVID-19; Vaccine Adverse Reaction; Side Effect; Inflammation; Pain; Mulberry; IL-17
MeSH Terms: conditions — COVID-19; Inflammation; Pain

STUDY DESIGN:
Intervention Model Description: Participants are divided into three groups, namely, the low dose group (10 ml), middle dose group (50 ml), and high dose group (100 ml).
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants are told that they would receive a cup of mulberry juice in which the volume is randomized, without knowing the exact dose range.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low volume mulberry juice (Experimental): 10 ml mulberry juice containing about 48 mg polyphenols
  Interventions: Dietary Supplement: Mulberry juice
- Middle volume mulberry juice (Experimental): 50 ml mulberry juice containing about 240 mg polyphenols
  Interventions: Dietary Supplement: Mulberry juice
- High volume mulberry juice (Experimental): 100 ml mulberry juice containing about 480 mg polyphenols
  Interventions: Dietary Supplement: Mulberry juice

INTERVENTIONS:
Dietary Supplement: Mulberry juice — Mulberry is a common macrophanerophyte that can be found in fields or farms. Mulberry fruits contain a large amount of anthocyanins and a relatively small amount of pro-anthocyanins. The plant is easy to grow and the fruit price is low compared with other types of plants producing anthocyanins, and thus a reliable source for anthocyanin supplements. Current laboratory evidence has shown that specific anthocyanins can reduce inflammation status, and potentially thrombosis. One of the enzymes inhibited by specific anthocyanins is cyclooxygenase which catalyzes the synthesis of prostanoids, including thromboxane and prostaglandins. Moreover, a critical study has shown that cyanidin 3-O-glucoside, the main anthocyanin in mulberry fruit, is an allosteric regulator of interleukin-17A.

SUMMARY:
Urgent vaccine development plus the characteristics of the coronavirus have caused the relatively more safety problems in COVID-19 vaccines than other classic vaccines and unavoidably raises more concerns among those who accept or consider to be vaccinated. Mulberry juice consists of a large amount of anthocyanin. The abnormally high interleukin-17A level is frequently seen in patients with inflammation status or diseases with inflammation features. Some specific anthocyanins can reduce cyclooxygenase and nitrogen oxide, and the pharmacological effect of the major anthocyanin in mulberry juice imitates that of interleukin-17A antagonists. These features make mulberry juice a potential crude material for reducing inflammation and pain induced by COVID-19 vaccinations. The investigators propose a randomized control trial to explore the dose-response effects of three different volumes of mulberry juice on the incidence and severity of COVID-19 induced side effects. The findings should be helpful for nutrition supplementation in COVID-19 vaccinations and may improve public coordination of COVID-19 vaccinations.

DETAILED DESCRIPTION:
Since the outbreak of Coronavirus Disease-2019 (COVID-19), the size of the infected population continues to expand, and the number of deaths due to the infection continues to climb. Massive vaccination has become the most critical measure to control the pandemic. Vaccination may cause side effects. Urgent vaccine development plus the characteristics of the coronavirus have caused the relatively more safety problems in COVID-19 vaccines than other classic vaccines and unavoidably raises more concerns among those who accept or consider to be vaccinated. Mulberry juice consists of a large amount of anthocyanin. The abnormally high interleukin-17A level is frequently seen in patients with inflammation status or diseases with inflammation features. Previous cell and animal studies have shown that some specific anthocyanins can reduce cyclooxygenase and nitrogen oxide, and the pharmacological effect of the major anthocyanin in mulberry juice imitates that of interleukin-17A antagonists. These features make mulberry juice a potential crude material for reducing inflammation and pain induced by COVID-19 vaccinations. The investigators propose a randomized control trial investigating the dose-response effects of three different volumes of mulberry juice on the incidence and severity of COVID-19 induced side effects and build up initial dose-response models for future reference in nutrition supplementation in COVID-19 vaccinations and improve public coordination of COVID-19 vaccinations.

ELIGIBILITY:
Inclusion Criteria:

* Concious
* Mentally capable
* Can comunicate using Mendalin or Taiwanese dialet
* Agree to join the current trial

Exclusion Criteria:

* Unable to read the google sheets
* dysphagia
* > 65 years

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2022-05-31 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Change of body temperature | Up to four days
  Daily body temperature of each participant is recorded to obtain serial temperatures including body temperature before vaccination (first day) and body temperatures after vaccination (second, third, and fourth day).
Number of participants with fever | Up to four days
  Event of 38 degrees celsius or above

SECONDARY OUTCOMES:
Number of participants with sign cluster 1 (multiple choices) | Up to three days
  Redness, swelling, pain, lump or mass, or rash and itching at the injection site; axillary swelling and tenderness at the injection arm; axillary swelling and tenderness at the non-injection arm; none
Number of participants with sign cluster 2 (multiple choices) | Up to three days
  Chills, headache, muscle pain, joint pain, fatigue, rash on the body, asthma or breathing difficulty, loss of appetite, nausea or vomiting, diarrhea, stomach ache, insomnia, or drownsiness; none

CONTACTS AND LOCATIONS:
Overall Officials: El-Wui Loh, PhD, Principal Investigator — Taipei Medical University Shuang Ho Hospital